CLINICAL TRIAL: NCT00115479
Title: KULeuven Intensive Insulin Therapy Study in Medical Intensive Care Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S18630; FWO grant number G.0278.03; KULeuven OT/03/56
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2005-06

CONDITIONS: Critical Illness
Keywords: critical illness; intensive care; outcome; insulin; blood glucose
MeSH Terms: conditions — Critical Illness; Insulin Resistance

INTERVENTIONS:
Drug: intensive insulin therapy to maintain normoglycemia

SUMMARY:
In a previous study, we showed that tight blood glucose control with insulin during intensive care reduced morbidity and mortality of surgical intensive care patients. Whether this intervention also improves prognosis of medical intensive care patients remains unknown. The current prospective, randomized, controlled study will assess the impact of intensive insulin therapy on the outcome of patients in a medical intensive care unit. On admission, patients will be randomly assigned to either strict normalization of blood glucose (80-110 mg/dl) with intensive insulin therapy or the conventional approach, in which insulin infusion is initiated only when blood glucose exceeds 215 mg/dl, to maintain blood glucose levels between 180 and 200 mg/dl.

DETAILED DESCRIPTION:
In a previous study, we showed that tight blood glucose control with insulin during intensive care reduced morbidity and mortality of surgical intensive care patients. Whether this intervention also improves prognosis of medical intensive care patients remains unknown. The current prospective, randomized, controlled study will assess the impact of intensive insulin therapy on the outcome of patients in a medical intensive care unit. On admission, patients will be randomly assigned to either strict normalization of blood glucose (80-110 mg/dl) with intensive insulin therapy or the conventional approach, in which insulin infusion is initiated only when blood glucose exceeds 215 mg/dl, to maintain blood glucose levels between 180 and 200 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to ICU and anticipated to require intensive care for at least a few days

Exclusion Criteria:

* Expected short ICU stay
* Therapy restricted upon admission
* Surgical ICU patients
* Other studies
* Below 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2002-03; Study Completion 2005-06

PRIMARY OUTCOMES:
mortality

SECONDARY OUTCOMES:
mechanical ventilatory support-dependency
stay in Intensive Care Unit (ICU)
stay in hospital
organ failure
morbidity
a long-term follow up is planned to take place 6 and 12 months after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Greet H Van den Berghe, MD, PhD, Principal Investigator — K.U.Leuven
Locations (1):
- Catholic University of Leuven, University Hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Result] Van den Berghe G, Wilmer A, Hermans G, Meersseman W, Wouters PJ, Milants I, Van Wijngaerden E, Bobbaers H, Bouillon R. Intensive insulin therapy in the medical ICU. N Engl J Med. 2006 Feb 2;354(5):449-61. doi: 10.1056/NEJMoa052521. PMID 16452557
- [Derived] Boonen E, Vervenne H, Meersseman P, Andrew R, Mortier L, Declercq PE, Vanwijngaerden YM, Spriet I, Wouters PJ, Vander Perre S, Langouche L, Vanhorebeek I, Walker BR, Van den Berghe G. Reduced cortisol metabolism during critical illness. N Engl J Med. 2013 Apr 18;368(16):1477-88. doi: 10.1056/NEJMoa1214969. Epub 2013 Mar 19. PMID 23506003
- [Derived] Langouche L, Vander Perre S, Frystyk J, Flyvbjerg A, Hansen TK, Van den Berghe G. Adiponectin, retinol-binding protein 4, and leptin in protracted critical illness of pulmonary origin. Crit Care. 2009;13(4):R112. doi: 10.1186/cc7956. Epub 2009 Jul 9. PMID 19589139